CLINICAL TRIAL: NCT04664049
Title: The Outcomes of NRICM101 on SARS-COV-2 (COVID-19) Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Research Institute of Chinese Medicine, Ministry of Health and Welfare (Other Government)
Responsible Party: Sponsor
Other Study IDs: NRICM101
Record Dates: First submitted 2020-12-04; First posted 2020-12-11 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: SARS-CoV-2; Covid 19
Keywords: NRICM101; Covid 19; SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NRICM101: Subjects who confirmed, suspected or prevented infected of COVID 19 disease and received dietary supplement NRICM101
  Interventions: Dietary Supplement: NRICM101

INTERVENTIONS:
Dietary Supplement: NRICM101 — Direction: Take 1 sachet 2-4 times daily directly or with 400cc water before or between meals
  Indication: Externally contracted seasonal epidemic
  Function: Relieving Exterior and Facilitating Lung, clear heat of lung, Wide chest and resolve phlegm

SUMMARY:
Traditional Chinese medicine is regarded as a dietary supplement in many countries around the world. Dietary supplement, NRICM101, has been available for people who diagnosed, suspected or prevented for coronavirus disease 2019 (COVID-19) in September 2020. It is expected to help people not to progress to severe illness, and reduce lung damage and mortality. The investigators gather the effects of people who taking NRICM101 using the Real-World Big Data Study and the network feedback information collection model. This study can be used as a reference for global prevention and control of coronavirus disease 2019 (COVID-19).

DETAILED DESCRIPTION:
The Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) is raging around the world. Because of its strong spread, variability, survivability, and invisibility, the number of infected people rise rapidly. On March 11, 2020, the WHO officially declared COVID-19 as a pandemic disease. As of October 3, 2020, the number of confirmed cases has exceeded 34 million, and the cumulative deaths have exceeded 1 million. There are still no drugs to treatment the coronavirus disease 2019 (COVID-19). Due to the mutation of virus rapidly, vaccine development cannot be completed in a short period of time. At the beginning of the infection outbreak, the governments of China and South Korea, adopted a cooperative of Chinese and Western medicine to treatment the coronavirus disease 2019 (COVID-19). In addition to the reported good clinical effects, Chinese medicine prescriptions have included in diagnosis and treatment guideline of these two countries.

Traditional Chinese medicine is regarded as a dietary supplement in many countries around the world. Dietary supplement, NRICM101, has been available for people who diagnosed, suspected or prevented for coronavirus disease 2019 (COVID-19) in September 2020. It is expected to help people not to progress to severe illness, and reduce lung damage and mortality. The investigators gather the effects of people who taking NRICM101 using the Real-World Big Data Study and the network feedback information collection model. This study can be used as a reference for global prevention and control of coronavirus disease 2019 (COVID-19).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who confirmed, suspected or prevented infected of COVID 19 disease and take dietary supplement NRICM101

Exclusion Criteria:

* Those who refuse to participate in observational research.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who confirmed, suspected or prevented infected of COVID 19 disease and take dietary supplement NRICM101
Sampling Method: Non-Probability Sample
Enrollment: 51000 (Estimated)
Dates: Start 2020-12-23 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
negative of COVID-19 test | 1 day to 2 months
  receive COVID 19 test and the result is negative
free of COVID 19 disease symptoms and signs | 1 day to 2 months
  free of COVID 19 disease symptoms and signs after took NRICM101

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Chang Su, MD, PhD, Principal Investigator — National Research Institute of Chinese Medicine, Ministry of Health and Welfare
Locations (1):
- National Research Institute of Chinese Medicine, Ministry of Health and Welfare, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided